CLINICAL TRIAL: NCT02563106
Title: A Double-Blind, Placebo-Controlled, Multicenter Study of SYN-004 Compared to Placebo for the Prevention of C.Diff in Patients With a Diagnosis of a Lower Respiratory Tract Infection
Brief Title: A Study of SYN-004 for the Prevention of C.Diff in Patients With a LRTI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theriva Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SB-2-004-005
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Clostridium Difficile; Clostridium Infections
MeSH Terms: conditions — Clostridium Infections | interventions — SYN-004

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SYN-004 (Experimental): SYN-004 150 mg
  Interventions: Drug: SYN-004
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYN-004
  Arms: SYN-004
Drug: Placebo
  Arms: Placebo

SUMMARY:
A Phase 2b Parallel-Group, Double-Blind, Placebo-Controlled, Multicenter Study of SYN-004 Compared to Placebo for the Prevention of Clostridium difficile Infection (CDI) in Hospitalized Patients receiving IV ceftriaxone with a Diagnosis of a Lower Respiratory Tract Infection (LRTI).

DETAILED DESCRIPTION:
This is a Phase 2b, randomized, double-blind, placebo controlled, parallel-group, multi-center proof-of-concept study to assess the potential of SYN-004 in the prevention of CDI and the unwanted side effects of IV antibiotic treatment in at risk patients who are hospitalized for LRTI and receiving IV ceftriaxone alone or in combination with a macrolide. Subjects will be 50 years or older. The entire duration of the study may be up to 59 days. All patients will be evaluated for the occurrence of CDI and AAD by testing according to local diagnostic standards and monitoring for diarrhea (3 or more unformed stools per 24 hour period).

ELIGIBILITY:
Inclusion Criteria:

* Expected minimum hospital stay of 5 days
* Expected ≥5 day course of intravenous (IV) ceftriaxone alone or in combination with a macrolide
* Clinical diagnosis of moderate to severe lower respiratory tract infection consisting of signs and symptoms of a lower respiratory tract infection and Pneumonia Severity Index (PSI/PORT) score for CAP of 90-130, inclusive. Evidence of a new or progressive infiltrate on chest x-ray is recommended.

Exclusion Criteria:

* Presence of a diarrheal illness within 72 hours prior to randomization
* Current treatment for CDAD or ongoing active CDI, as evidenced by clinical signs of diarrhea along with the presence of toxin A and/or B (or their respective genes, tcdA and/or tcdB) of C. difficile in the stool
* Number of previous CDAD episodes >1 within 12 weeks of randomization and no C. difficile infection (CDI) within 4 weeks of randomization
* Use of antibiotics within 1 month of start of study drug except for the current illness.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2015-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kaleko, MD, Study Director — Synthetic Biologics
Locations (43):
- United States (6):
  - Synthetic Biologics Investigational Site, Little Rock, Arkansas
  - Synthetic Biologics Investigational Site, Torrance, California
  - Synthetic Biologics Investigational Site, DeLand, Florida
  - Synthetic Biologics Investigational Site, Będzin, Louisiana
  - Synthetic Biologics Investigational Site, Debrecen, Louisiana
  - Synthetic Biologics Investigational SIte, Natchitoches, Louisiana
- Bulgaria (8):
  - Synthetic Biologics Investigational Site, Gabrovo
  - Synthetic Biologics Investigational Site, Kyustendil
  - Synthetic Biologics Investigational Site, Lovech
  - Synthetic Biologics Investigational Site, Multiple Locations
  - Synthetic Biologics Investigational Site, Rousse
  - Synthetic Biologics Investigational Site, Sevlievo
  - Synthetic Biologics Investigational Site, Sofia
  - Synthetic Biologics Investigational Site, Targovishte
- Canada (2):
  - Synthetic Biologics Investigational Site, Sherbrooke
  - Synthetic Biologics Investigational Site, Toronto
- Hungary (3):
  - Synthetic Biologics Investigational Site, Balassagyarmat
  - Synthetic Biologics Investigational Site, Budapest
  - Synthetic Biologics Investigational Site, Veszprém
- Poland (11):
  - Synthetic Biologics Investigational Site, Bialystok
  - Synthetic Biologics Investigational Site, Bochnia
  - Synthetic Biologics Investigational Site, Bydgoszcz
  - Synthetic Biologics Investigational Site, Chodzież
  - Synthetic Biologics Investigational Site, Lodz
  - Synthetic Biologics Investigational Site, Oława
  - Synthetic Biologics Investigational Site, Pomorskie
  - Synthetic Biologics Investigational Site, Siedlce
  - Synthetic Biologics Investigational Site, Tarnów
  - SyntheticBiologics Investigational Site, Tychy
  - Synthetic Biologics Investigational Site, Warszawice
- Romania (7):
  - Synthetic Biologics Investigational Site, Arad
  - Synthetic Biologics Investigational Site, Brasov
  - Synthetic Biologics Investigational SIte, Bucharest
  - Synthetic Biologics Investigational Site, Cluj-Napoca
  - Synthetic Biologics Investigational Site, Oradea
  - Synthetic Biologics Investigational Site, Otopeni
  - Synthetic Biologics Investigational Site, Timișoara
- Serbia (6):
  - Synthetic Biologics Investigational Site, Belgrade
  - Synthetic Biologics Investigational Site, Čačak
  - Synthetic Biologics Investigational Site, Gornji Matejevac
  - Synthetic Biologics Investigational Site, Kragujevac
  - Synthetic Biologics Investigational Site, Novi Sad
  - Synthetic Biologics Investigational Site, Užice

REFERENCES:
- [Derived] Kokai-Kun JF, Roberts T, Coughlin O, Le C, Whalen H, Stevenson R, Wacher VJ, Sliman J. Use of ribaxamase (SYN-004), a beta-lactamase, to prevent Clostridium difficile infection in beta-lactam-treated patients: a double-blind, phase 2b, randomised placebo-controlled trial. Lancet Infect Dis. 2019 May;19(5):487-496. doi: 10.1016/S1473-3099(18)30731-X. Epub 2019 Mar 15. PMID 30885591

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (no active drug)
Period: Overall Study
Arm/Group | SYN-004 | Placebo
Started | 206 | 207
Completed | 172 | 178
Not Completed | 34 | 29
Not completed — Withdrawal by Subject | 7 | 8
Not completed — Adverse Event | 17 | 15
Not completed — Protocol Violation | 1 | 0
Not completed — Use of non-permitted concurrent therapy | 1 | 2
Not completed — Lost to Follow-up | 3 | 2
Not completed — Physician Decision | 3 | 1
Not completed — Other reason - not specified | 2 | 1

BASELINE CHARACTERISTICS:
Population: One subject in the placebo group was randomized but never dosed. The subject withdrew consent prior to dosing, therefore they are not included in the analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | SYN-004 | Placebo | Total
Number analyzed (Participants) | 206 | 206 | 412
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (9.37) | 69.7 (9.37) | 69.2 (9.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 80 | 153
  Male | 133 | 126 | 259
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 206 | 205 | 411
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Europe | 203 | 201 | 404
  North America | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Clostridium Difficile Infection at 4- Weeks of Follow-up.
Description: Percentage of subjects with CDI, based on the protocol definition of CDI (defined as 3 or more unformed stools per 24 hour period and a stool sample being positive for C. difficile toxin A and/or B [or their respective genes, tcdA and/or tcdB], based on the clinical site local laboratory results) from Day 1 to the 4-week Follow-up Visit in the SYN-004 treatment group compared to the placebo group, imputing early termination without CDI as not being treatment failures.
Time Frame: Day 1 to the 4 week Follow-up Visit.
Population: The Modified Intent-to-Treat (mITT) analysis set included randomized subjects who received at least 1dose of study drug. Number of subjects with CDI, imputing early termination without CDI as not being treatment failures.
Measure: Count of Participants; unit: Participants
Arm/Group | SYN-004 | Placebo
Number analyzed (Participants) | 206 | 206
Participants | 2 | 7
Statistical Analysis 1: Comparison: SYN-004 vs Placebo; The Modified Intent-to-Treat (mITT) analysis set included randomized subjects who received at least 1 dose of study drug. Number of subjects with CDI, imputing early termination without CDI as not being treatment failures; Test type: Other — The analysis of the primary endpoint was based on the mITT analysis set. Per-protocol and worse case analyses were performed as sensitivity analyses.The P-value was based on a one-sided z-test for the comparison of the treatment difference between the SYN-004 group and the Placebo group; p = 0.045, z-test — Study was designed to provide 80% power to detect treatment effect with one-sided alpha = 0.05 on the primary endpoint. Based on the pre-specified z-test the one-sided P=0.045; 1-sided P=0.045; Relative Risk Reduction (%) = 71.4, 95% CI 2-sided [-35.9 to 94.0] — Relative Risk Reduction in SYN-004 group compared to Placebo group

ADVERSE EVENTS:
Time Frame: 6 weeks.
Description: The "Total" reported in the "Other (Not Including Serious) Adverse Events (AEs) Section" for SYN-004 and Placebo indicate the total number of AEs. The number of subjects "Affected" by those AEs is 42 for SYN-004 and 46 for Placebo.
  The frequency threshold of 1% for non-serious adverse events is reported as the # of subjects w/ AEs (excluding Serious Adverse Events (SAEs)) in each group, based on # of subjects w/ AEs >1% in the SYN-004 group & the corresponding AE categories for Placebo group.
Arm/Group | SYN-004 | Placebo
All-Cause Mortality (participants affected / at risk) | 11/206 | 5/206
Serious Adverse Events (participants affected / at risk) | 33/206 | 21/206
Other Adverse Events (participants affected / at risk) | 59/206 | 59/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SYN-004 (N=206) | Placebo (N=206)
Anemia of Chronic Disease (Blood and lymphatic system disorders) | 0 | 1
Iron Deficiency Anemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 2
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Bronchopneumonia (Infections and infestations) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Empyema (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 5
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
International normalised ratio abnormal (Investigations) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Chronic lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYN-004 (N=206) | Placebo (N=206)
Hypertension (Vascular disorders) | 7 (7) | 10 (13)
Constipation (Gastrointestinal disorders) | 7 (10) | 6 (7)
Insomnia (Nervous system disorders) | 4 (4) | 9 (9)
Headache (Nervous system disorders) | 5 (5) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 11 (11)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5)
Atrial Fibrillation (Cardiac disorders) | 3 (3) | 2 (2)
Oral Candidiasis (Infections and infestations) | 3 (3) | 3 (3)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
A safety assessment conducted by an independent third party to evaluate SAEs and fatal events confirmed that they were related to the subjects' underlying health, medical history, and comorbidities and not to study drug administration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators do not see trial results ahead of public disclosure unless it is under CDA. Investigators will not be allowed to publish or disclose any study results prior to sponsor communicating it to the public.